CLINICAL TRIAL: NCT02339753
Title: Pharmacokinetic Study of Carboplatin in Pediatric Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Korean Society of Pediatric Hematology Oncology (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH_carboplatinPK
Record Dates: First submitted 2015-01-02; First posted 2015-01-15 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Pediatric Solid Tumor
MeSH Terms: interventions — Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin-treatment arm (Experimental): Arm description : Carboplatin intravenous administration once daily for 3 to 4 days
  * Topotecan + Thiotepa + Carboplatin : carboplatin 500mg/m2/day, for 3 days
  * MEC for 2nd PBSCT : carboplatin 350 mg/m2/day, for 4 days
  * MEC for other solid tumor : carboplatin 400 mg/m2/day, for 4 days
  * MEC + MIBG Tx for 2nd PBSCT (neuroblastoma) : carboplatin 300 mg/m2/day, for 4 days
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin — Blood sampling will be done at the time before administration (0hr pre-dose), 1hr, 2hr, 5hr for pharmacokinetic study.
  Other Names: Neoplatin

SUMMARY:
Carboplatin is widely used for conditioning regimens of autologous hematopoietic stem cell transplantation for pediatric solid tumor, but the pharmacokinetics has not been evaluated in pediatric stem cell transplantation before. As carboplatin have renal toxicity, the pharmacokinetic study of carboplatin would help the safe and effective administration of carboplatin for transplantation patients. Especially, the dose of carboplatin is higher at conditioning chemotherapy, resulting in higher toxicity.

Carboplatin is a drug mostly excreted by kidney, and the dose of carboplatin is recommended according to the body surface area and kidney function, represented by glomerular filtration rate. After analyzing the pharmacokinetics of carboplatin, analyses will also be done for the methods to determine the appropriate carboplatin dose.

DETAILED DESCRIPTION:
Purpose

1. Primary objective: To evaluate the pharmacokinetics of carboplatin in pediatric HSCT patients.
2. Secondary objective: To evaluate the toxicity of HSCTs using carboplatin as the conditioning regimen. To compare the pharmacokinetics of carboplatin in adults and children.

Eligibility Inclusion criteria

1. Patients who undergo HSCT with conditioning regimen including carboplatin. 2. Age under 19 years. 3. Performance status: ECOG 0-2. 4. Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases.

1. Heart: a shortening fraction > 30% and ejection fraction > 45%.
2. Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal.
3. Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.

5. Patients must lack any active viral infections or active fungal infection. 6. Patients (or one of parents if patients age < 19) should sign informed consent.

Exclusion criteria

1. Pregnant or nursing women.
2. Malignant or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
3. Psychiatric disorder that would preclude compliance.
4. If the clinician decides that there is a condition improper for the clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who undergo HSCT with conditioning regimen including carboplatin. 2. Age under 19 years. 3. Performance status: ECOG 0-2. 4. Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases.

1. Heart: a shortening fraction > 30% and ejection fraction > 45%.
2. Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal.
3. Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.

5. Patients must lack any active viral infections or active fungal infection. 6. Patients (or one of parents if patients age < 19) should sign informed consent.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Malignant or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
3. Psychiatric disorder that would preclude compliance.
4. If the clinician decides that there is a condition improper for the clinical study.

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve (AUC) of carboplatin at the first and last administration day | From the start of first dose carboplatin administration to 5 hours from the last administration

SECONDARY OUTCOMES:
Number of participants with adverse events after HSCT using carboplatin as the conditioning regimen | From the start of carboplatin administration to 100 days from hematopoietic stem cell transplantation
  Especially, kidney function will be focused.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Shin, MD, PhD, Principal Investigator — Department of Pediatrics, Cancer Research Institute, Seoul National University College of Medicine, Seoul, Korea
Locations (1):
- Seoul National University Hospital, Seoul, South Korea